CLINICAL TRIAL: NCT06618365
Title: Oral or Intra Muscular Vitamin D2 Vs Oral or Intra Muscular Vitamin D3 in Treatment of Vitamin D Deficiency.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr Hassan Saqr, Senior Consultant, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-18-036
Record Dates: First submitted 2024-09-08; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Endocrinology
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: prospective randomized intervention using open label randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Vitamin D2 50000 units per tablet (Experimental): They will take one tablet weekly.
  Interventions: Drug: Vitamin D Deficiency
- Group 2: Vitamin D2 300000 units Intramuscular injection (Experimental): They will have one injection every 6 weeks initially.
  Interventions: Drug: Vitamin D Deficiency
- Group 3: Vitamin D3 50000 units tablet (Experimental): They will take one tablet weekly.
  Interventions: Drug: Vitamin D Deficiency
- Group 4: Vitamin D3 300000 units Intramuscular injection (Experimental): They will have one injection every 6 weeks initially.
  Interventions: Drug: Vitamin D Deficiency

INTERVENTIONS:
Drug: Vitamin D Deficiency — The first phase will involve studying 4 groups with the outcome (percentage of patients attaining Vitamin D levels >30ng/ml) at 3 months to show the superiority of any of the groups. Vitamin D levels will be checked at baseline then 6 and 12 weeks. The second phase will include only patients who achieve the target level above 30ng/ml after the first phase and will be randomized to receive either oral Vitamin D2 or oral Vitamin D3 every 2, 3 or 4 weeks for another 3 months.
  For patients that achieved normal level in phase 1, we will keep a maintenance dose of the oral Vitamin D for 2 groups with 3 sub-groups under each.

SUMMARY:
The main purpose of this research is to find out if there is any difference between treating vitamin D deficiency with oral vitamin D3 or I.M vitamin D2. The second aim of this research is to confirm the superiority of Vitamin D3 over Vitamin D2 in treating vitamin D deficiency. Additional useful information in this research is to find out the best recommended maintenance dose of vitamin D and formula by having regular follow up of treated individuals once their serum vitamin D level reach the recommended normal serum level.

DETAILED DESCRIPTION:
In a systemic review, it was found that treating individuals who have vitamin D deficiency with vitamin D3 rather than vitamin D2 would be a better option. Vitamin D3 is superior in treating Vitamin D deficiency according to this systemic review. However, this systemic review raised a question of comparing oral to I.M treatment of vitamin D deficiency and no Data was available to support either treatment above the other.

The main purpose of this research is to find out if there is any difference between treating vitamin D deficiency with oral vitamin D3 or I.M vitamin D2. The second aim of this research is to confirm the superiority of Vitamin D3 over Vitamin D2 in treating vitamin D deficiency. Additional useful information in this research is to find out the best recommended maintenance dose of vitamin D and formula by having regular follow up of treated individuals once their serum vitamin D level reach the recommended normal serum level.

The research will involve 100 patients between the age of 20-50 years old. They will be divided into 4 groups. Each group will have either oral or I.M vitamin D2 or oral or I.M vitamin D3. The oral doses will be 50000 international units to be taken weekly and the I.M doses will be of 300000 international units which will be taken once every 6 weeks. Vitamin D level will be checked once every 4 weeks. The initial expected duration of the first phase of the research will be about 6-12 weeks which will give us a good orientation to answer the main and the second questions. Then the follow up may take up to another 6 months to check the maintenance dose of the best recommended oral or I.M treatment of bolus doses in certain intervals as initial trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years
* Basal Vit D level should be between 10-18 ng/ml for phase 1 and between 30-50 ng/ml for phase 2

Exclusion Criteria:

* Pregnant Women
* history of renal implant or renal impairment of eGFR less than 60%
* Abnormal Liver function test
* patients with inflammatory bowel disease or of history of bariatric surgery

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Is oral Vitamin D3 superior to I.M Vitamin D2 in treating vitamin D deficiency? | 3 months from the administration of first dose
  The primary outcome will be evaluated after 3 months from administration of the first dose for each subject to assess the serum level of vitamin D is attained. If a subject has reached normal Vitamin D serum level, they are qualified for phase 2 of the study.

SECONDARY OUTCOMES:
Confirming superiority of oral Vitamin D3 over oral Vitamin D2 | 3 months after administration of the first dose.
  The secondary outcome of confirming the superiority of oral Vitamin D3 over oral Vitamin D2 in treating vitamin D deficiency will be evaluated after a subject has completed 3 months since the administration of the first dose.
to compare the treatment of vitamin D deficiency by using intramuscular injection of vitamin D3 or Vitamin D2 | 3 months after administration of the first dose.
  The third outcome also to compare the treatment of vitamin D deficiency by using intramuscular injection of vitamin D3 or Vitamin D2 and establish if there is any treatment is superior to another if we are using the intramuscular injections.

OTHER OUTCOMES:
evaluating recommended maintenance dose in certain time intervals of oral vitamin D3 and Vitamin D2 | 24 weeks from initial baseline
  The fourth outcome of evaluating recommended maintenance dose in certain time intervals of oral vitamin D3 and Vitamin D2.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
This was not intended initially, and the consent form does not include any clause for the participants to request sharing their data with other researchers.